CLINICAL TRIAL: NCT06098079
Title: A Phase IV Study to Assess the Effect of Naltrexone Hydrochloride Extended Release (ER) and Bupropion Hydrochloride ER Combination (Contrave®/Mysimba®) on the Occurrence of Major Adverse Cardiovascular Events
Brief Title: Effect of Naltrexone Hydrochloride ER and Bupropion Hydrochloride ER Combination (Contrave®/Mysimba®) on Major Adverse Cardiovascular Events (MACE)
Acronym: INFORMUS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Currax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NB-CVOT3
Record Dates: First submitted 2023-10-13; First posted 2023-10-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor will be blinded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naltrexone/Bupropion (NB) (Active Comparator): Patients will be randomly assigned to NB (naltrexone 8 mg and bupropion 90 mg) extended-release oral tablet.
  Interventions: Drug: Naltrexone-Bupropion (NB) Combination
- Placebo (Placebo Comparator): Patients will be randomly assigned to placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone-Bupropion (NB) Combination — A total daily dosage of two NB 8 mg/90 mg tablets twice daily (32 mg/360 mg) is reached at the start of Week 4.
  Arms: Naltrexone/Bupropion (NB)
Drug: Placebo — A total daily dosage of two placebo tablets twice daily (in an identical, non-medicine containing tablet) is reached at the start of Week 4.
  Arms: Placebo

SUMMARY:
A randomized, double-blinded, placebo controlled study intended to capture cardiovascular outcomes during real-world use of naltrexone/bupropion (NB).

DETAILED DESCRIPTION:
This multi-center, prospective, randomized, pragmatic, double-blinded study has been designed to capture cardiovascular (CV) outcomes during the real-world use of NB after initial randomization. The aim of the study is to assess whether patients receiving treatment with NB are at an elevated risk of experiencing MACE compared with patients receiving placebo. Both patient groups will also be counselled to lose weight via a reduced-calorie diet and increased physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥18 years at screening
2. Able to understand the key components of the study, as described in the written informed consent document, and willing and able to provide written informed consent
3. BMI ≥30 kg/m2 (obese) or ≥27 kg/m2 (overweight) in the presence of at least 1 weight-related comorbidity (eg, hypertension, type 2 diabetes mellitus, or dyslipidemia)
4. At increased risk of adverse cardiovascular outcomes:

   In the opinion of the investigator, has a high likelihood of cardiovascular disease with at least 1 of the following:
   * History of documented MI >90 days prior to screening
   * History of coronary revascularization (ie, coronary artery bypass graft surgery, stent placement, percutaneous transluminal coronary angioplasty, or laser atherectomy) >90 days prior to screening
   * History of carotid or peripheral revascularization (ie, carotid endarterectomy, lower extremity atherosclerotic disease atherectomy, repair of abdominal aorta aneurysm, femoral or popliteal bypass) >90 days prior to screening
   * Angina with ischemic changes (resting echocardiogram (ECHO), ECG changes on a graded exercise test (GXT), or positive cardiac imaging study)
   * Ankle brachial index <0.9 (by simple palpation) within prior 2 years or

   Type 2 diabetes mellitus with at least 2 of the following:
   * Hypertension (controlled with or without pharmacotherapy at <145/95 mmHg)
   * Dyslipidemia requiring pharmacotherapy
   * Documented low HDL cholesterol (<50 mg/dL in women or <40 mg/dL in men) within the prior 12 months
   * Current tobacco smoker
5. Patients who have completed a washout (2-weeks or 5 half-lives, whichever is longer) of the prohibited concomitant medication(s) at screening
6. Subject willing to comply with daily completion of an eDiary using a mobile smartphone application

Exclusion Criteria:

1. Using prescription medications, other than Contrave/Mysimba, or surgical or medical device interventions for weight loss
2. History of MI or stroke within 90 days prior to screening
3. Uncontrolled hypertension, defined as systolic BP ≥160 mmHg and/or >100 mmHg diastolic BP on the average of 3 seated BP measurements after the patient has been at rest for at least 5 minutes
4. Meets any of the following criteria:

   * Confirmed end-stage renal disease (ie, a degree of kidney failure severe enough to require dialysis or kidney transplantation for survival characterized by a severe reduction in glomerular filtration rate [<15 mL/minute/1.73 m2] and other manifestations including increased serum creatinine),
   * Severe hepatic impairment (Child-Pugh score 10 to 15 [Class C]),
   * Hemodynamic instability, including patients with severe heart failure (New York Heart Association Class IV)
5. Seizure disorders or history of seizures, not including subjects with a history of pediatric febrile seizures
6. Use of other bupropion-containing products (including but not limited to Wellbutrin, Wellbutrin SR, Wellbutrin XL, and Aplenzin)
7. Active anorexia nervosa or bulimia
8. Chronic opioid or opiate agonist (eg, methadone) or partial agonists (eg, buprenorphine) use, or acute opioid withdrawal or has a positive urine drug result for opioids at screening
9. Undergoing abrupt discontinuation of alcohol, benzodiazepines, barbiturates, and antiepileptic drugs
10. Concomitant administration of MAOIs. This also includes use of reversible MAOIs, such as linezolid or intravenous methylene blue. At least 14 days should elapse between discontinuation of MAOIs and initiation of treatment with Contrave/Mysimba.
11. Subject has any disease or condition, or use of any pharmacological agent to treat the disease/condition, that, in the opinion of the investigator, would contraindicate study participation
12. Known allergy to bupropion, naltrexone, or any other component of Contrave/Mysimba
13. Pregnant or nursing
14. Known life-threatening arrythmias, including Brugada syndrome
15. Participation in any other concurrent investigational trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8600 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Cardiovascular Death | Treatment initiation through 1 year following treatment termination.
  Occurrence of cardiovascular death in number of study patients receiving NB compared with number of study patients receiving placebo.
Occurrence of Non-fatal Myocardial Infarction (MI) | Treatment initiation through 1 year following treatment termination.
  Occurrence of MI in number of study patients receiving NB compared with number of study patients receiving placebo. MI will be identified using current standard diagnostic criteria, such as the 2017 Cardiovascular and Stroke Endpoints Definitions for Clinical Trials.
Occurrence of Non-fatal Stroke | Treatment initiation through 1 year following treatment termination.
  Occurrence of non-fatal stroke in number of study patients receiving NB compared with number of study patients receiving placebo. Stroke will be identified using current standard diagnostic criteria, such as the 2017 Cardiovascular and Stroke Endpoints Definitions for Clinical Trials.

SECONDARY OUTCOMES:
Comparative Rates of Cardiovascular Death | Treatment initiation through 1 year following treatment termination.
  Comparative rates of cardiovascular death between number of study patients receiving NB compared to number of study patients receiving placebo.
Comparative Rates of Non-fatal Myocardial Infarction (MI) | Treatment initiation through 1 year following treatment termination.
  Comparative rates of non-fatal MI between number of study patients receiving NB compared to number of study patients receiving placebo.
Comparative Rates of Non-fatal Stroke | Treatment initiation through 1 year following treatment termination.
  Comparative rates of non-fatal stroke between number of study patients receiving NB compared to number of study patients receiving placebo.

CONTACTS AND LOCATIONS:
Locations (140):
- United States (140):
  - TrialMed Birmingham (DRS), Birmingham, Alabama
  - Accel Research Sites Network, Birmingham, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - AMR Mobile, Mobile, Alabama
  - Velocity Clinical Research, Mobile, Mobile, Alabama
  - Sun City Research, Glendale, Arizona
  - Cardiovascular Consultants/NextStage Clinical Research, Glendale, Arizona
  - Desert Clinical Research, Mesa, Arizona
  - Velocity Clinical Research, Phoenix, Phoenix, Arizona
  - Fiel Family & Sports Medicine CCT Research, Tempe, Arizona
  - Synexus Clinical Research US; Inc., Tucson, Arizona
  - Velocity Clinical Research, Gardena, Anderson, California
  - Velocity Clinical Research, Chula Vista, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Chemidox Clinical Trials Inc., Lancaster, California
  - Long Beach Clinical Trials, Long Beach, California
  - Velocity Clinical Research, Los Angeles, California
  - Valley Vitality Ventures, Manteca, California
  - National Institute of Clinical Research, Inc., Pomona, California
  - Velocity Clinical Research, San Bernardino, San Bernardino, California
  - Velocity Clinical Research at Coastal Heart Medical Group, Santa Ana, California
  - Velocity Clinical Research of Santa Ana, Santa Ana, California
  - Velocity Clinical Research, Van Nuys, Van Nuys, California
  - Providere Research, West Covina, California
  - Velocity Clinical Research, Denver, Englewood, Colorado
  - ABMED Clinical Research, Cape Coral, Florida
  - LMG Research, Coral Gables, Florida
  - JY Research Institute, Cutler Bay, Florida
  - Delray Physician Center, Delray Beach, Florida
  - D&H Doral Research Center, Doral, Florida
  - Accel Research Sites Network - Edgewater, Edgewater, Florida
  - Velocity Clinical Research (New Smyrna Beach), Edgewater, Florida
  - IMRC Fort Lauderdale, Fort Lauderdale, Florida
  - Southwest General Healthcare Center, Fort Myers, Florida
  - G+C Research Group, Hialeah, Florida
  - Qway Research, Hialeah, Florida
  - Conveinent Medical Research, Hialeah, Florida
  - Ilumina Medical Research, Kissimmee, Florida
  - Altus Research, Lake Worth, Florida
  - D&H Pompano Research Center, LLC, Margate, Florida
  - Optimal Research, LLC. - Melbourne, Melbourne, Florida
  - Advanced Clinical Research, Miami, Florida
  - Medical Research Center Westchester, Miami, Florida
  - Century Research, Miami, Florida
  - ITB Research, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Janus Clinical Research, Miami, Florida
  - Miami Beach Clinical Research, Miami Beach, Florida
  - Innovia Research Center, Miramar, Florida
  - Healix Clinical Research, New Smyrna Beach, Florida
  - Biscayne Clinical Research Inc, North Miami, Florida
  - IMRC At Palmetto Bay, Palmetto Bay, Florida
  - New Horizons Research, Palmetto Bay, Florida
  - Best Choice Medical and Research Services, Pembroke Pines, Florida
  - Bolanos Clnical Research, Pembroke Pines, Florida
  - Cordova Research Institute, Sweetwater, Florida
  - D&H Tamarac Research Center, LLC, Tamarac, Florida
  - Synexus Clinical Research US, Inc. - The Villages, The Villages, Florida
  - Advanced Clinical Research Atlanta, Atlanta, Georgia
  - Clincept Clinical Research, Columbus, Georgia
  - Accel Research Sites (ARSN) - Neurostudies, Decatur, Georgia
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - NextStage Clinical Research-Chicago, Glen Ellyn, Illinois
  - JAELEX Research, Round Lake Beach, Illinois
  - Indiana Medical Research Institute, Merriville, Indiana
  - Velocity Clinical Research, Valparaiso, Indiana
  - Velocity Clinical Research, Sioux City, Iowa
  - AMR - El Dorado, El Dorado, Kansas
  - Velocity Clinical Research, Kansas City, Kansas City, Kansas
  - AMR Wichita West, Wichita, Kansas
  - AMR Wichita East, Wichita, Kansas
  - Wichita Surgical Specialists, Wichita, Kansas
  - Velocity Clinical Research, Baton Rouge, Louisiana
  - Tandem Clinical Research, Covington, Louisiana
  - Velocity Clinical Research, Covington, Louisiana
  - Velocity Clinical Research, Lafayette, Louisiana
  - AMR New Orleans, New Orleans, Louisiana
  - Velocity Clinical Research, New Orleans, New Orleans, Louisiana
  - Velocity Clinical Research, Slidell, Louisiana
  - Regenerative Orthopedics and Sports Medicine- NextStage Clinical Research, North Bethesda, Maryland
  - Praveen K Gupta, MD/Avacare, Rockville, Maryland
  - Velocity Clinical Research, Rockville, Rockville, Maryland
  - Activmed Practices and Research, Inc, Methuen, Massachusetts
  - Dearborn Cardiology, Dearborn, Michigan
  - Velocity Clinical Research, Gulfport, Mississippi
  - Clay Platte Family Medicine, Kansas City, Missouri
  - St. Louis Medical Professionals/CCT Research, St Louis, Missouri
  - Velocity Clinical Research, Grand Island, Grand Island, Nebraska
  - Velocity Clinical Research at Pioneer Heart Institute, Lincoln, Nebraska
  - Velocity Clinical Research, Lincoln, Nebraska
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Meridian Clinical Research - Velocity, Omaha, Nebraska
  - Midwest Regional Health Services, Omaha, Nebraska
  - Avacare, Las Vegas, Nevada
  - Santa Rosa Urgent Care Primary Care/CCT Research, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - ActivMed Practices and Research, Portsmouth, New Hampshire
  - Velocity Clinical Research, Albuquerque, New Mexico
  - Axces Research Group, Santa Fe, New Mexico
  - Velocity Clinical Research, Binghamton, New York
  - Synexus Clinical Research US, Inc. - New York, New York, New York
  - Velocity Clinical Research, Vestal, New York
  - Velocity Clinical Research, Durham, Durham, North Carolina
  - Velocity Clinical Research, Beachwood, Ohio
  - Velocity Clinical Research, Mt. Auburn, Cincinnati, Ohio
  - Velocity Clinical Research, Cincinnati, Cincinnati, Ohio
  - Velocity Clinical Research, Cincinnati, Ohio
  - NexGen Research, Lima, Ohio
  - NextStage Clinical Research - Tulsa, Tulsa, Oklahoma
  - Velocity Clinical Research, Grants Pass, Grants Pass, Oregon
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Hatboro Medical Associates/Avacare Research, Horsham, Pennsylvania
  - Mercado Medical Practice/CCT Research, Philadelphia, Pennsylvania
  - Velocity Clinical Research (Providence), East Greenwich, Rhode Island
  - Velocity Clinical Research, Anderson, South Carolina
  - Velocity Clinical Research, Charleston, South Carolina
  - Velocity Clinical Research, Columbia, South Carolina
  - Velocity Clinical Research, Gaffney, South Carolina
  - Velocity Clinical Research, Greenville, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Velocity Clinical Research, Spartanburg, Spartanburg, South Carolina
  - Velocity Clinical Research, Union, Union, South Carolina
  - Velocity Clinical Research, Abilene, Abilene, Texas
  - Optimal Research, LLC. - Austin, Austin, Texas
  - Velocity Clinical Research, Austin, Texas
  - Advanced Cardiovascular Specialists/NextStage Clinical Research, Beaumont, Texas
  - HDH Research, Houston, Texas
  - All-American Orthopedics-NextStage Clinical Research, Houston, Texas
  - NextStage Clinical Research-Lubbock/SWAT Surgical Associates-NextStage Clinical Research, Lubbock, Texas
  - NextStage Clinical Research-Port Arthur/Gulf Coast Cardiology, Port Arthur, Texas
  - Synexus Clinical Research US; Inc., San Antonio, Texas
  - Olympus Clinical Research, Sugarland, Texas
  - Waco Cardiology Consultants, Waco, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Velocity Clinical Research, Hampton, Hampton, Virginia
  - AMR Norfolk, Norfolk, Virginia
  - Velocity Clinical Research, Suffolk, VA, Suffolk, Virginia
  - Evergreen Surgical, Eau Claire, Wisconsin